CLINICAL TRIAL: NCT04335006
Title: A Multicentre, Open-parallel, Randomized, Controlled Phase Ⅲ Study Comparing Carelizumab Plus Nab-paclitaxel and Apatinib, Carelizumab Plus Nab-paclitaxel, and Nab-paclitaxel in Patients With Unresectable Locally Advanced or Metastatic Triple Negative Breast Cancer.
Brief Title: A Phase 3 Study Comparing Carelizumab Plus Nab-paclitaxel and Apatinib, Carelizumab Plus Nab-paclitaxel, and Nab-paclitaxel in Patients With Advanced Triple Negative Breast Cancer.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor R & D Strategy Adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-III-318
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
Keywords: SHR-1210; PD-1
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — camrelizumab; 130-nm albumin-bound paclitaxel; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental A (Experimental): Subjects receive Carelizumab in combination with Nab-paclitaxel plus Apatinib,each 4-week cycle
  Interventions: Drug: Carelizumab; Drug: Nab-paclitaxel; Drug: Apatinib
- Experimental B (Experimental): Subjects receive Carelizumab in combination with Nab-paclitaxel,each 4-week cycle
  Interventions: Drug: Carelizumab; Drug: Nab-paclitaxel
- Comparator C (Active Comparator): Subjects receive nab-paclitaxel intravenously each 4-week cycle.
  Interventions: Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Carelizumab — Participants receive SHR-1210 intravenously (IV)
  Other Names: SHR-1210
  Arms: Experimental A; Experimental B
Drug: Nab-paclitaxel — administered intravenously every 4-week cycle
Drug: Apatinib — administered orally every 4-week cycle
  Arms: Experimental A

SUMMARY:
This randomized, open-label phase 3 study will evaluate the safety and efficacy of Carelizumab (an engineered anti-programmed death-ligand 1 [PD-1] antibody) in combination with Nab-paclitaxel and Apatinib, carelizumab plus nab-paclitaxel, and Nab-paclitaxel in Patients with Unresectable Locally Advanced or Metastatic Triple Negative Breast Cancer. Participants will be randomized in a 1:1:1 ratio to Arm A (Carelizumab + Nab-paclitaxel + Apatinib), Arm B (Carelizumab + Nab-paclitaxel), or Arm C (Nab-paclitaxel).

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0-1.
* Expected lifetime of not less than three months
* Metastatic or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression)
* Cancer stage: locally advanced or metastatic breast cancer; Locally advanced breast cancer not amenable to radical resection.
* No prior systemic antitumor therapy for metastatic triple-negative breast cancer.
* Adequate hematologic and organ function
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)

Exclusion Criteria:

* Known central nervous system (CNS) disease.
* Previously received anti-VEGFR small molecule tyrosine kinase inhibitors or anti-PD-1/PD-L1 antibody.
* A history of bleeding, any serious bleeding events.
* Uncontrolled pleural effusion, pericardial effusion.
* Malignancies other than TNBC within 5 years prior to randomisation, or ascites requiring recurrent drainage procedures
* History of interstitial pneumonitis.
* Severe chronic or active infections in need of systemic antibacterial, antifungal, or antiviral treatment, including TB, etc.
* Prior allogeneic stem cell or solid organ transplantation.
* History of autoimmune disease
* Active hepatitis B or hepatitis C
* Pregnancy or lactation.
* Peripheral neuropathy grade ≥2.
* Participants with poor blood pressure control;
* Myocardial infarction incident within 6 months prior to randomisation;
* Treatment with systemic immunostimulatory agents within 4 weeks prior to randomisation
* Treatment with systemic immunosuppressive medications within 2 weeks prior to randomisation

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Randomisation to the first occurrence of disease progression or death (through the end of study, approximately 42 months)
  Progression-free survival (PFS) as determined by the IRC according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) in PD-L1 positive / ITT population

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 42 months
  Progression Free Survival (PFS) as determined by the investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1) in PD-L1 positive/ITT population
Overall Survival (OS) in PD-L1 positive/ITT population | Up to approximately 42 months
Objective response rate (ORR) in the PD-L1-positive/ITT population | Up to approximately 42 months
Clinical benefit rate (CBR), defined as the proportion of patients with a CR or a PR or stable disease as determined by the investigator according to RECIST 1.1 | Up to approximately 42 months
Percentage of Participants with Adverse Events (AEs) | Up to approximately 42 months
Serum concentration of SHR-1210 and plasma concentration of apatinib | Up to approximately 42 months
Proportion of anti-SHR-1210 antibody (ADA) and neutralizing antibody (Nab) formed during the study from baseline | Up to approximately 42 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No